CLINICAL TRIAL: NCT01373086
Title: A Multi-center, Randomized, Double-blind, Placebo and Active Controlled, Parallel Group, Proof-of-concept Study to Evaluate the Efficacy and Safety of LFF269 Compared to Placebo After Treatment in Subjects With Essential Hypertension
Brief Title: LFF269 Compared to Placebo After Treatment in Subjects With Essential Hypertension
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLFF269X2201
Record Dates: First submitted 2011-05-24; First posted 2011-06-14 (Estimated); Last update posted 2020-12-17 (Actual); Status verified 2012-11

CONDITIONS: Hypertension
Keywords: Hypertension,; mild hypertension,; moderate hypertension,; high blood pressure,; uncomplicated hypertension.
MeSH Terms: conditions — Hypertension | interventions — Eplerenone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- LFF269 low dose (Experimental): LFF269 low dose + Matching Placebo to Eplerenone 50mg during 4 week double blind period
  Interventions: Drug: LFF269; Drug: Placebo
- LFF269 high dose (Experimental): LFF269 high dose + Matching Placebo to Eplerenone 50mg
  Interventions: Drug: LFF269; Drug: Placebo
- Eplerenone (Active Comparator): Eplerenone 50mg twice daily + matching placebo of LFF269
  Interventions: Drug: Eplerenone; Drug: Placebo
- Placebo (Placebo Comparator): Placebo of LFF269 high dose + Placebo of Eplerenone 50 mg
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LFF269
  Arms: LFF269 high dose; LFF269 low dose
Drug: Eplerenone
  Arms: Eplerenone
Drug: Placebo

SUMMARY:
This study will assess the efficacy and safety of LFF269 compared to placebo after treatment in subjects with essential hypertension.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female (post-menopausal or surgically sterile).
2. Age from 18 to 75 years inclusive.
3. Subjects with mild-to-moderate uncomplicated essential hypertension, with (not more than 2 in combination) or without prior treatment.
4. Subjects must weigh at least 50 kg to participate in the study, and must have a body mass index (BMI) within the range of 18 - 36 kg/m2.

Exclusion Criteria:

1. History or evidence of a secondary form of hypertension,
2. History of cardiovascular disease. Type 1 or type 2 diabetes mellitus.
3. Clinically significant valvular heart disease.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2011-05; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in mean 24-hour systolic blood pressure (SBP) as measured by ambulatory blood pressure monitoring (ABPM) after 4 weeks treatment | Baseline, week 4

SECONDARY OUTCOMES:
Change from baseline in mean 24-hour diastolic blood pressure (DBP) as measured by ABPM after 4 weeks of treatment | Baseline, week 4
Change from baseline in mean 24-hour SBP and DBP as measured by ABPM after 4 weeks treatment | Baseline, week 4
Percentage of patients experiencing adverse events during the study as measure of safety and tolerability | 4 weeks
  Adverse events will be reported as percentage of patients with total adverse events, serious adverse events and death.
Change from baseline in mean sitting SBP and DBP after 4 weeks treatment | Baseline, week 4
Percentage of patients achieving a successful BP response (> placebo) and BP control (SBP < 140 mmHg at trough) | 4 weeks
change from baseline in mean daytime and mean nighttime SBP and DBP as measured by ABPM after 4 weeks treatment | Baseline, week 4
Pharmacokinetics of LFF269: Plasma concentrations of LFF269 | pre dose & 6 hours post study drug dose

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (11):
- United States (11):
  - Advanced Clinical Research Institute-Phase I, Anaheim, California
  - Comprehensive Phase I, Fort Myers, Florida
  - Comprehensive Phase One®,, Miramar, Florida
  - Comprehensive NeuroScience, St. Petersburg, Florida
  - Clinical Research Atlanta, Stockbridge, Georgia
  - Clinical Research Advantage/ Prairie Fields Family Medicine, PC, Fremont, Nebraska
  - Internal Medicine Physicians, Omaha, Nebraska
  - ICON Developmental Solutions, Omaha, Nebraska
  - Clinical Research Advantage/ Aloha Medical, Las Vegas, Nevada
  - ICON Development Solutions,, San Antonio, Texas
  - Comprehensive Clinical Development NW, Inc., Tacoma, Washington

REFERENCES:
- See also: Results for CLFF269X2201 from the Novartis Clinical Trials website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=7184